CLINICAL TRIAL: NCT02953132
Title: A Randomised, Double-Blind, Placebo-Controlled, First-Time-in-Human Study to Determine the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of MT-4129 in Healthy Subjects; Including the Effect of Gender and Age on the Pharmacokinetics of a Single Dose of MT-4129 in Healthy Subjects
Brief Title: A Clinical Study to See How the Study Drug MT-4129 is Taken up by the Body in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MT-4129-E01
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Healthy

ARMS (2):
- Single ascending dose, MT-4129 or Placebo (Experimental)
  Interventions: Drug: MT-4129; Drug: Placebo
- Multiple ascending dose, MT-4129 or Placebo (Experimental)
  Interventions: Drug: MT-4129; Drug: Placebo

INTERVENTIONS:
Drug: MT-4129
Drug: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of ascending single and multiple oral doses of MT-4129 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and free from clinically significant illness or disease
* Male or female subjects aged 18 to 55 years or elderly male subjects aged ≥65
* A body weight of ≥60 kg for males and ≥50 kg for females, and a body mass index ranging from 18 to 30 kg/m2

Exclusion Criteria:

* Participated in more than three clinical studies involving administration of an IMP in the previous year, or any study within 12 weeks
* Clinically significant endocrine, thyroid, hepatic, respiratory, gastro intestinal, neurological, renal, cardiovascular disease, or history of any significant psychiatric/psychotic illness disorder
* Clinically relevant abnormal medical history, physical findings or laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as measured by incidence and severity of adverse events | Up to Day 14
Safety and Tolerability as measured by vital signs | Up to Day 14
Safety and Tolerability as measured by ECG | Up to Day 14
Safety and Tolerability as measured by clinical laboratory assessments | Up to Day 14
Safety and Tolerability as measured by Hormone assessments | Up to Day 10
Safety and Tolerability as measured by physical examination | Up to Day 14

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of MT-4129 | Up to Day 10
Measured time of maximum observed plasma concentration (tmax) of MT-4129 | Up to Day 10
Apparent terminal elimination half-life (t1/2) of MT-4129 | Up to Day 10
AUC from time zero to 24 hours post-dose (AUC0-24) of MT-4129 | Up to Day 8
AUC from time zero to 48 hours post-dose (AUC0-48) of MT-4129 | Up to Day 9
AUC from time zero to 72 hours post-dose (AUC0-72) of MT-4129 | Up to Day 10
AUC from time zero to infinity (AUC0-∞) of MT-4129 | Up to Day 10
AUC from time zero to the last measurable concentration (AUC0-last) of MT-4129 | Up to Day 10
AUC over the dosing interval (AUC0-t) of MT-4129 | Up to Day 10
Terminal elimination rate constant (Kel) of MT-4129 | Up to Day 10
Mean residence time (MRT) of MT-4129 | Up to Day 10
Apparent volume of distribution during terminal phase after oral administration (Vz/F) of MT-4129 | Up to Day 10
Apparent volume of distribution at steady state (Vss/F) of MT-4129 | Up to Day 10
Apparent oral clearance (CL/F) of MT-4129 | Up to Day 10
Urinary excreted amount of test compound (Ae) of MT-4129 | Up to Day 10
Urinary excreted amount of test compound expressed as a percentage of the dose administered (Ae%) of MT-4129 | Up to Day 10
Renal clearance (CLR) of MT-4129 | Up to Day 10
Plasma aldosterone | Up to Day 10
Serum cortisol | Up to Day 10
Plasma steroid hormones | Up to Day 10
Urinary aldosterone | Up to Day 10
Urinary cortisol | Up to Day 10
Urinary sodium | Up to Day 10
Urine potassium | Up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Pharmaceutical Research Associates (PRA) Health Sciences, City Name, Netherlands